CLINICAL TRIAL: NCT02778360
Title: Effectiveness of a Personalized Neurofeedback Training Device (ADHD@Home) as Compared With Methylphenidate in the Treatment of Children and Adolescents With Attention-Deficit/Hyperactivity Disorder: A Multicentre Randomized Clinical Study
Brief Title: Effectiveness of a Personalized Neurofeedback Training Device (ADHD@Home) in Attention-Deficit/Hyperactivity Disorder
Acronym: Newrofeed
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mensia Technologies SA (Industry)
Collaborators: European Union H2020 SME Instrument (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Newrofeed
Record Dates: First submitted 2016-05-12; First posted 2016-05-19 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Attention Deficit-Hyperactivity Disorder
Keywords: Attention deficit; Neurofeedback; ADHD; Methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neurofeedback NFT (Experimental): Neurofeedback Training based on real time electroencephalography (EEG) signal. The patient is trained to modulate his brain activity thanks to a tablet installed with serious game.
  Initiation/Discovery period during 21 days: initiation and discovery sessions Treatment period during 9 weeks: 36 training sessions at home
  Interventions: Device: Neurofeedback NFT
- Methylphenidate MPH (Active Comparator): Methylphenidate long acting preparation.
  Open titration protocol during 21 days: 10 mg/day as a start until optimal dose is reached (maximum dose: 60 mg/day).
  Treatment period during 9 weeks: optimal dose with MPH LA 10 and 30 mg (dose range: 10 mg/day to 60 mg/day).
  Interventions: Drug: Methylphenidate MPH

INTERVENTIONS:
Device: Neurofeedback NFT — The ADHD@Home Device is composed of a software for NF Training deployed on a Windows tablet, and connected to an EEG headset and an amplifier.
  The training is personalized according to patient's characteristics.
  Other Names: Neurofeedback training; ADHD@Home
  Arms: Neurofeedback NFT
Drug: Methylphenidate MPH — Drug prescribed with a first titration period until an optimal dose.
  Other Names: Methylphenidate long acting; Medikinet retard
  Arms: Methylphenidate MPH

SUMMARY:
The main objective of the study is to demonstrate the non-inferiority of the personalized Neurofeedback Training device versus Methylphenidate in the treatment of children and adolescents with Attention-Deficit/Hyperactivity Disorder.

DETAILED DESCRIPTION:
The main objective of the present study is to demonstrate the non-inferiority of the personalized Neurofeedback Training device ADHD@Home versus Methylphenidate in the treatment of children and adolescents with Attention-Deficit/Hyperactivity Disorder.

Furthermore, it is aimed to learn more about the mechanisms underlying NeuroFeedback.

The study is prospective, multicentric (9 centres), randomised, reference drug-controlled.

ADHD@Home is a neuromarkerTM-based personalized medicine device to treat children suffering from Attention Deficit Hyperactivity Disorders (ADHD) with Neurofeedback Training (NFT) based on real time electroencephalography (EEG) signal.

Neurofeedback Training is based on direct training of brain function, by which the brain learns to function more efficiently. For each session of the ADHD@Home solution, the child is trained to modulate his brain activity in a serious game, which is a real-time metaphor of the EEG biomarker that needs to be 'normalized', following a typical operant learning process.

ELIGIBILITY:
Inclusion Criteria:

* Children or adolescents (male or female) aged 7-13 years
* ADHD diagnosis positive with Kiddie-Sads
* ADHD RS IV >6 for attention, with or without hyperactivity
* Patient having already had corrective actions for ADHD (formal and informal educational support, psychoeducation, psychotherapy, occupational therapy remediation, at-school programs and remediations)
* Signature of inform consent form by parent and child
* Wireless internet connection at home

Exclusion Criteria:

* ADHD hyperactive/Impulsive without inattention component
* Established diagnosis of epilepsy or other neurological disorders
* Severe and/or uncontrolled psychiatric disorder other than ADHD diagnosed with Kiddie-Sads such as autism, schizophrenia, severe generalized anxiety disorder, major depression or severe tics
* Patient with comorbid disorder requiring psychoactive medication other than ADHD medication
* Patient having already been treated with psycho-active drug (MPH and others) or EEG-NF for ADHD in the last 6 months, or more than 4 weeks more than 6 months ago
* Unable to use the solution (tablet use and/or headset set-up and/or understanding instructions) according to the investigator
* Absence of wireless internet connection at home
* Medical disorder requiring systemic chronic medication with confounding psychoactive effects
* IQ < 80 using the 3 subtest form of the WASI or the WISC
* Plans to move requiring centre change during the next 6 months
* Plans to start other ADHD treatment, including psychotherapy, cognitive behaviour training in the next 6 months
* Patient with chronic medical illness such as seizure, cardiac disorders, untreated thyroid disease or glaucoma (contra-indication for treatment with MPH)
* Significant suicidal risk based on clinical opinion
* Patient with prescribed dietary interventions
* Patient with a known hypersensitivity to one of the ingredients of the investigational products

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 179 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Change from Day 0 at Day 90 of the total score of the ADHD RS IV (Attention Deficit Hyperactivity Disorder Rating Scale IV) | 3 times (Day 0, Day 60, Day 90)
  ADHD RS IV (Attention Deficit Hyperactivity Disorder Rating Scale IV): total score assessed by the clinician

SECONDARY OUTCOMES:
ADHD RS IV Inattention and Hyperactivity Sub-Scores | 3 times (Day 0, Day 60, Day 90)
  ADHD RS IV (Attention Deficit Hyperactivity Disorder Rating Scale IV): Inattention and Hyperactivity sub-scores assessed by the clinician
Clinical responders | 1 time (Day 90)
  Clinical responders are subjects who will present a decrease of the total clinician ADHD RS score of more or equal to 25%
Parents ADHD RS IV Total, Inattention and Hyperactivity Scores | 3 times (Day 0, Day 60, Day 90)
  ADHD RS IV (Attention Deficit Hyperactivity Disorder Rating Scale IV): Total, Inattention and Hyperactivity scores assessed by the parents
Teacher ADHD RS IV Total, Inattention and Hyperactivity Scores | 2 times (Day 0, Day 90)
  ADHD RS IV (Attention Deficit Hyperactivity Disorder Rating Scale IV): Total, Inattention and Hyperactivity scores assessed by the teacher
Clinical Global Impression (severity) (CGI-S) | 7 times (Day 0, Day 7, Day 14, Day 21, Day 28, Day 60, Day 90)
  Severity of the illness assessed by the clinician
Clinical Global Impression (improvement) (CGI-I) | 6 times (Day 7, Day 14, Day 21, Day 28, Day 60, Day 90)
  Improvement of the patient's condition assessed by the clinician
Behavior Rating Inventory of Executive Function (BRIEF) | 2 times (Day 0, Day 90)
  Executive Function Tests by the Behavior Rating Inventory of Executive Function (BRIEF)
Conners Continuous Performance Test 3rd Edition (Conners CPT 3) | 2 times (Day 0, Day 90)
  Conners Continuous Performance Test 3rd Edition
Strengths and Difficulties Questionnaire (SDQ) | 2 times (Day 0, Day 90)
  Behaviour assessment by the parents and the teacher with the Strengths and Difficulties Questionnaire
quantitative Electro-Encephalogram (qEEG) | 3 times (Day 0, Day 60, Day 90)
  Quantitative electroencephalogram to assess EEG biomarkers, progress in brain modulation
Columbia suicide severity rating scale (C-SSRS) | 7 times (Day 0, Day 7, Day 14, Day 21, Day 28, Day 60, Day 90)
  Columbia suicide severity rating scale
Sleep Disturbance Scale for Children (SDSC) | 7 times (Day 0, Day 7, Day 14, Day 21, Day 28, Day 60, Day 90)
  Sleep Disturbance Scale for Children
Pediatric adverse event rating scale (PAERS) | 7 times (Day 0, Day 7, Day 14, Day 21, Day 28, Day 60, Day 90)
  Pediatric adverse event rating scale
Physical examination | 1 time (Day 0)
  Physical examination will include assessments of height, weight, cardiac frequency, cardiac exam and blood pressure.
  Investigator will question the parents about the cardiac history of the family and on individual risk factors. If a risk factor is detected, the patient will be addressed to a cardiologist for an electrocardiogram (ECG).
Medical/surgical history | 1 time (Day 0)
  Assessment especially related to the eligibility criteria
Concomitant treatments collection | 7 times (Day 0, Day 7, Day 14, Day 21, Day 28, Day 60, Day 90)
  All the treatments taken during the participation will be collected (trade name, indication, dose, onset/end dates).
  The use of concomitant medications will be summarized by therapeutic class.
Adverse events collection | 6 times (Day 7, Day 14, Day 21, Day 28, Day 60, Day 90)
  All the adverse events occurred during the participation will be collected until resolution or stabilization (description/symptoms, onset/end dates, frequency, intensity, evolution, causality to treatment attributed, seriousness).
  All adverse events will be described in each arm. A comparison will be done, especially concerning number and percentage of patients who experienced at least one adverse event (on the whole and by system/organ), at least one adverse event leading to discontinue the treatment, and at least one serious adverse event.
Child Health and Illness Profile, Child Edition (CHIP-CE) | 2 times (Day 0, Day 90)
  Measure of the quality of life by the parents with the CHIP-CE parents report form

CONTACTS AND LOCATIONS:
Overall Officials: Michel Du Peloux, PhD, Study Director — Mensia Technologies; Diane Purper-Ouakil, MD/PhD, Principal Investigator — CHRU Montpellier
Locations (12):
- Belgium (2):
  - PSY Pluriel Centre europeen de psychologie medicale, Brussels
  - Hôpital Erasme - Cliniques universitaires de Bruxelles, Brussels
- France (5):
  - Centre Hospitalier Charles Perrens, Bordeaux
  - CHRU de Lille - Hôpital Fontan - Service de psychiatrie de l'enfant et de l'adolescent, Lille
  - Clinique LAUTREAMONT, Lille
  - Hospice Civil de Lyon - Hôpital Neurologique Service de Neuro-Psychiatrie de l'Enfant, Lyon
  - CHRU Montpellier, Montpellier
- Germany (2):
  - Universitätklinikum Erlangen, Erlangen, Bavaria
  - Medical faculty of Mannheim/Heidelberg university, Mannheim
- Puerta de Hierro Hospital - Department of Psychiatry, Madrid, Spain
- Switzerland (2):
  - Clinique des Grangettes, Geneva
  - Psychiatric Hospital, University of Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Purper-Ouakil D, Blasco-Fontecilla H, Ros T, Acquaviva E, Banaschewski T, Baumeister S, Bousquet E, Bussalb A, Delhaye M, Delorme R, Drechsler R, Goujon A, Hage A, Kaiser A, Mayaud L, Mechler K, Menache C, Revol O, Tagwerker F, Walitza S, Werling AM, Bioulac S, Brandeis D. Personalized at-home neurofeedback compared to long-acting methylphenidate in children with ADHD: NEWROFEED, a European randomized noninferiority trial. J Child Psychol Psychiatry. 2022 Feb;63(2):187-198. doi: 10.1111/jcpp.13462. Epub 2021 Jun 24. PMID 34165190
- [Derived] Bioulac S, Purper-Ouakil D, Ros T, Blasco-Fontecilla H, Prats M, Mayaud L, Brandeis D. Personalized at-home neurofeedback compared with long-acting methylphenidate in an european non-inferiority randomized trial in children with ADHD. BMC Psychiatry. 2019 Aug 1;19(1):237. doi: 10.1186/s12888-019-2218-0. PMID 31370811
- See also: Opinons on NFT for ADHD — http://www.mensiatech.com/neurofeedbackinadhd/